CLINICAL TRIAL: NCT02294240
Title: Effect of Energy Dense Biscuits in Under Nourished Pregnant Women on Birth Weight of Their Newborns in a Low Income Peri-urban Setting of Karachi; a Community Based Randomized Interventional Study
Brief Title: Effect of Energy Dense Biscuits in Undernourished Women on Birth Weight of Their Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aga Khan University (Other)
Collaborators: English Biscuit Manufacturers (Unknown)
Responsible Party: Principal Investigator, Dr Faraz Naz Qamar, Assistant professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PED 3009
Record Dates: First submitted 2014-11-05; First posted 2014-11-19 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Birth Weight
Keywords: Pregnant, malnourished, energy dense biscuits, low birth weight
MeSH Terms: conditions — Birth Weight; Malnutrition | interventions — Flour; Oils; Iron; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm One (Experimental): Energy dense biscuits will be provided throughout pregnancy after enrolment
  Interventions: Dietary Supplement: Energy dense biscuits
- Arm Two (Placebo Comparator): Wheat Flour,oil, iron and folic acid will be provided fortnightly throughout pregnancy after enrolment
  Interventions: Other: Wheat Flour, oil, iron & Folic acid

INTERVENTIONS:
Dietary Supplement: Energy dense biscuits — Energy dense biscuits will be provided
  Arms: Arm One
Other: Wheat Flour, oil, iron & Folic acid — Wheat flour, oil, iron and folic acid will be provided
  Arms: Arm Two

SUMMARY:
A nutrition trial which is based on the evidence that multivitamins & micro nutrients provided during pregnancy in malnourished women will improve neonatal birth weight. There will be two arms. Arm one will provide energy dense biscuits to pregnant women with BMI <20 & gestational age less than 14 weeks. The other arm with same criteria will be provided with wheat flour, oil, iron & folic acid. Neonatal birth weight is the primary outcome of interest but maternal weight gain, maternal hemoglobin & ferritin levels and palatability of biscuits will also be assessed.

DETAILED DESCRIPTION:
It has been realized that micronutrient deficiencies are a major determinant of intra-uterine growth retardation (IUGR) so multiple trials using micronutrient supplementation during pregnancy have been done & shown a positive effect on birth weight.UNICEF/WHO/United Nations University(UNU) designed a new multiple micro nutrient supplement for pregnant and lactating women-the UNICEF/WHO/UNU international multiple micro nutrient preparation (UNIMMAP)-that provides the Recommended Dietary Allowance (RDA) of 15 vitamins and minerals. The benefit of this supplementation over routinely prescribed iron and folic supplementation has been proven in multiple trials. Evidence has shown reduction in low birth newborns.

This randomized controlled trial will compare the effect of calories and multiple micro nutrients provided in energy dense biscuits manufactured by EBM to malnourished pregnant women seen by AKU's Department of Paediatrics and Child Health at their Ali Akbar Shah Goth and Ibrahim Hyderi, compared to food supplementation ration of wheat and oil, plus iron and folic acid tablet supplementation.

Arm 1: Dietary supplementation with EBM biscuits containing multiple vitamins and calcium in the recommended allowance (RDA) for pregnant women Arm 2: Supplementation with Wheat flour and oil, iron and folic acid All undernourished pregnant females identified before 14 weeks of gestation through our surveillance system will be offered enrollment.

First contact: First meeting will be on enrollment. Patients will be randomized into any one of the arm. After randomization Weight, height, MUAC and BMI will be recorded. Samples for Ferritin & hemoglobin will be drawn. In Arm 1 participant will be supplied with energy dense biscuits while in arm 2 will be provided with Wheat flour and oil after every two weeks.

End of each trimester: In second(20-22 week) & third trimester(33-35 week) weight, MUAC & BMI will be recorded. Supplementation will be given according to the Arm. Samples will also be drawn for Ferritin & hemoglobin on third visit. Also at the third trimester visit palatability, accessibility and compliance with biscuits will be assessed by filling a preformed questionnaire.

Follow up of the newborn: Follow up of the newborn will be done within 48 hours. Length, weight, fronto-occipital circumference and MUAC will be recorded.

ELIGIBILITY:
Inclusion Criteria:

All pregnant females with gestational age ≤14 weeks and Body mass index(BMI) <18.5

Exclusion Criteria:

Pregnant females with underlying chronic illness (cardiovascular disease, diabetes, renal disease, and hypertension)

Pregnant females with history of multiple abortions ( two or more abortions)

Pregnant females identified as having twin/triplet pregnancies

Pregnant females not consenting to participate

Pregnant females who are already enrolled in any other study that may interfere with the results of this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Neonatal birth weight | within 48 hours of birth
  Newborns will be captured within 48 hours of their birth and their birthweight will be measured

SECONDARY OUTCOMES:
Maternal weight gain | on enrolment,20-22 week, 33-35 week of gestation
  Maternal weight gain will be assessed by checking maternal weight on all three visits
Maternal Hemoglobin and Ferritin | On enrollment and last visit (33-35 weeks of gestation)
  Maternal Hemoglobin and Ferritin will be checked by drawing blood on enrollment and on 33-35 weeks of gestation
Palatability, acceptability, and compliance of the biscuits | On last visit (33-35 weeks of gestation)
  Palatability, acceptability, and compliance of the biscuits by filling a preformed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Farah N Qamar, Principal Investigator — Aga Khan University
Locations (2):
- Pakistan (2):
  - Ali Akbar Shah, Karachi, Sindh
  - Ibrahim Hyderi, Karachi, Sindh

REFERENCES:
- [Background] de Onis M, Blossner M, Villar J. Levels and patterns of intrauterine growth retardation in developing countries. Eur J Clin Nutr. 1998 Jan;52 Suppl 1:S5-15. PMID 9511014
- [Background] Kawai K, Spiegelman D, Shankar AH, Fawzi WW. Maternal multiple micronutrient supplementation and pregnancy outcomes in developing countries: meta-analysis and meta-regression. Bull World Health Organ. 2011 Jun 1;89(6):402-411B. doi: 10.2471/BLT.10.083758. Epub 2011 Mar 21. PMID 21673856
- [Background] Roberfroid D, Huybregts L, Lanou H, Henry MC, Meda N, Menten J, Kolsteren P; MISAME Study Group. Effects of maternal multiple micronutrient supplementation on fetal growth: a double-blind randomized controlled trial in rural Burkina Faso. Am J Clin Nutr. 2008 Nov;88(5):1330-40. doi: 10.3945/ajcn.2008.26296. PMID 18996870
- [Background] Berghella V. Prevention of recurrent fetal growth restriction. Obstet Gynecol. 2007 Oct;110(4):904-12. doi: 10.1097/01.AOG.0000267203.55718.aa. PMID 17906027
- [Background] Ramakrishnan U, Grant FK, Goldenberg T, Bui V, Imdad A, Bhutta ZA. Effect of multiple micronutrient supplementation on pregnancy and infant outcomes: a systematic review. Paediatr Perinat Epidemiol. 2012 Jul;26 Suppl 1:153-67. doi: 10.1111/j.1365-3016.2012.01276.x. PMID 22742608
- [Background] Osrin D, Vaidya A, Shrestha Y, Baniya RB, Manandhar DS, Adhikari RK, Filteau S, Tomkins A, Costello AM. Effects of antenatal multiple micronutrient supplementation on birthweight and gestational duration in Nepal: double-blind, randomised controlled trial. Lancet. 2005 Mar 12-18;365(9463):955-62. doi: 10.1016/S0140-6736(05)71084-9. PMID 15766997
- [Background] Gupta P, Ray M, Dua T, Radhakrishnan G, Kumar R, Sachdev HP. Multimicronutrient supplementation for undernourished pregnant women and the birth size of their offspring: a double-blind, randomized, placebo-controlled trial. Arch Pediatr Adolesc Med. 2007 Jan;161(1):58-64. doi: 10.1001/archpedi.161.1.58. PMID 17199068
- [Background] Jehan I, Harris H, Salat S, Zeb A, Mobeen N, Pasha O, McClure EM, Moore J, Wright LL, Goldenberg RL. Neonatal mortality, risk factors and causes: a prospective population-based cohort study in urban Pakistan. Bull World Health Organ. 2009 Feb;87(2):130-8. doi: 10.2471/blt.08.050963. PMID 19274365
- [Background] Imdad A, Bhutta ZA. Effect of balanced protein energy supplementation during pregnancy on birth outcomes. BMC Public Health. 2011 Apr 13;11 Suppl 3(Suppl 3):S17. doi: 10.1186/1471-2458-11-S3-S17. PMID 21501434
- [Background] Kramer MS, Kakuma R. Energy and protein intake in pregnancy. Cochrane Database Syst Rev. 2003;(4):CD000032. doi: 10.1002/14651858.CD000032. PMID 14583907